CLINICAL TRIAL: NCT03672526
Title: Use of Compuflo in Pediatric Anesthesia: Monitoring of Injection Pressure of Local Anesthetics in Children
Brief Title: Monitoring of Injection Pressure During Regional Anesthesia in Pediatric Patient
Acronym: COMPUFLO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: decision of the principal investigator
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL17_0399
Record Dates: First submitted 2018-09-11; First posted 2018-09-14 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Locoregional Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- device compuflo (Experimental)
  Interventions: Device: measure of injection pressure by compuflo

INTERVENTIONS:
Device: measure of injection pressure by compuflo — injection pressure mesured by Compuflo

SUMMARY:
A low injection pressure is one of the safety elements to check the correct position of the needle during regional anesthesia. Subjective assessment of pressure during manual injection of local anesthetic is most commonly used. In adults, the monitoring of the injection pressure has already been evaluated and makes it possible to objectify the pressure of the injection pressure. This is possible thanks to a device named Compuflo. No study has measured injection pressures during a regional anesthesia in children. The main objective is to control the injection pressures exercised in daily clinical practice during pediatric regional anesthesia with the Compuflo. Regional anesthesia will be proposed and explained during the anesthesia consultation. The procedure will be performed according to the habits of the anesthesiologist in charge of the patient. Only the addition of the Local Anesthetic Injection Pressure monitoring (Compuflo) to the needle changes the usual setup.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the usual practice using Compuflo, allowing the continuous measurement of the injection pressure of the local anesthetic at the needle level. On the day of the surgery, an anesthesiologist "operator" will realize the echo-guided regional anesthesia, qualifying aloud every injection realized (site or compartment of injection, and volume injected). An "observer" anesthesiologist will note the demographic data (age and weight), then the material data (minimum stimulation intensity, type and size of needles and syringes used), and finally he will note the maximum pressure levels reached during the injections performed.

ELIGIBILITY:
Inclusion Criteria:

* Minor patient (0-16 years old) with consent of the major legal representative
* Affiliated to the social security
* Informed written consent, notification on the anesthesia sheet

Exclusion Criteria:

* Patient over 16 years old
* Patient under tutorship / curatorship
* Young girl with known or suspected ongoing pregnancy
* Known allergy to local anesthetics
* Hemostatic disorder
* Local infection at the puncture site

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
injection pressure (injection pressure measured by Compuflo) | up to 24 hours (during the ALR)
  injection pressure measured by Compuflo

SECONDARY OUTCOMES:
Pressure values compared to the threshold value used in adults of 15 Psi | up to 24 hours (during the ALR)
  Pressure values compared to the threshold value used in adults of 15 Psi
Pressure values according to the different types of material used | up to 24 hours (during the ALR)
  Pressure values according to the different types of material used
Pressure values in the different infiltrated compartments | up to 24 hours (during the ALR)
  Pressure values in the different infiltrated compartments
Pressure values according to the age of the child | up to 24 hours (during the ALR)
  Pressure values according to the age of the child
Number and ratio of involuntary intra-neural injections | up to 24 hours (during the ALR)
  Number and ratio of involuntary intra-neural injections
Number and ratio of secondary paresthesias | up to 24 hours (during the ALR)
  Number and ratio of secondary paresthesias

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hertz L, Sola C, Pico J, Aros J, Scott C, Pirat P, Choquet O, Bringuier S, Dadure C. Objective real-time epidural pressure measurement using the CompuFlo(R) device, a mono-center observational study. Anaesth Crit Care Pain Med. 2025 Aug;44(4):101530. doi: 10.1016/j.accpm.2025.101530. Epub 2025 May 1. PMID 40318853